CLINICAL TRIAL: NCT06295107
Title: The Influence of Spasticity on Reliability of Range of Movement Measurements for Knee and Ankle in a Pediatric Population With Cerebral Palsy
Brief Title: Reliability of Range of Movement Measurements in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Olof Lindén, Consultant pediatric orthopedic surgeon, Region Skane
Other Study IDs: 2023-00195-01
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy; Movement Disorders in Children
Keywords: Cerebral palsy; Children; pROM; Goniometer; Spasticity; Reliability
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Spastic leg: Children with spastic hemiplegic cerebral palsy.
  Interventions: Diagnostic Test: Ankle Passive Range of Movement (pROM); Diagnostic Test: Knee Passive Range of Movement (pROM)
- Non spastic leg: Children with spastic hemiplegic cerebral palsy.
  Interventions: Diagnostic Test: Ankle Passive Range of Movement (pROM); Diagnostic Test: Knee Passive Range of Movement (pROM)

INTERVENTIONS:
Diagnostic Test: Ankle Passive Range of Movement (pROM) — Ankel and knee pROM measurements.
Diagnostic Test: Knee Passive Range of Movement (pROM) — Ankel and knee pROM measurements.

SUMMARY:
The aim is to investigate the inter-rater reliability of passive range of motion (pROM) measurement with goniometer of knee extension and ankle dorsiflexion for children with unilateral spastic cerebral palsy (USCP) and secondary to explore to what extent spasticity influences the reliability.

DETAILED DESCRIPTION:
Scientific question The aim is to investigate the inter-rater reliability of passive range of motion (pROM) measurement with goniometer of knee extension and ankle dorsiflexion for children with unilateral spastic cerebral palsy (USCP) and secondary to explore to what extent spasticity influences the reliability.

Overview of the field Evaluating joint mobility is commonly used and important for physicians and physiotherapists assessing and treating children with cerebral palsy, to early detect occurrence of joint contracture. The primarily used method to measure joint pROM is to use a manual goniometer, even if techniques using a smartphone or other electronic device has been demonstrated (Herrero et al. 2011, Ferriero et al. 2013, Hancock et al. 2018). Previous studies indicate that traditional goniometry is usually reliable both for ankle and knee both in individuals with and without spastic muscles (Brosseau et al. 2001, Allington et al. 2002, McWhirk et al. 2006, Konor et al. 2012) even if some authors indicate that there is a considerable variability among children with spasticity (McDowell et al. 2000).

To our knowledge no earlier study has investigated children with hemiplegic cerebral palsy to evaluate the influence of spasticity on pROM measurements. The idea is to use the child as its own control having both a spastic and a non spastic limb.

Project description

Participants Almost all children with cerebral palsy in Sweden are linked to a local habilitation unit where regular assessments are made by the child's physiotherapist. Information from the national quality registry and follow-up program for individuals with cerebral palsy (CPUP) indicates that there are approximately 140 children with unilateral spastic cerebral palsy (USCP) in Skåne. Families and children (age 2 - 17 years) with USCP linked to habilitation units in Skåne will be asked to participate in the study trough written letter and/or by phone call. When applicable this will be part of the child´s regular and planned assessment. Children with other diagnoses than USCP will be excluded. Children with surgery on the lower extremity within the last year or botox administration to the lower extremity within the last 3 month will also be excluded.

Methods The child will be assessed during one session of around 30-60 min. ROM measurements of knee extension and ankle dorsiflexion will be made on each child's both legs by two investigators with a standard two axis goniometer used in regular practice. The goniometer consists of two 20 cm arms attached in one end by a node and with a grade scale. The CPUP manual describes standardized patient positions and goniometer arm position for ROM in different joints.

For popliteal angle the child is positioned supine with the measured legs hip flexed to 90 degree while the other leg is fixed in extended position. The node of the goniometer is positioned lateral over the knee joint, the fixed arm aligned with femur and pointing towards the greater trochanter, the moving arm is held parallel to the anterior margin of tibia and pointing to the lateral malleolus.

Knee extension is examined with the child in supine position and extended knee, the node of the goniometer is positioned lateral over the knee joint center of rotation, the fixed arm aligned with femur and pointing towards the greater trochanter, the moving arm is held parallel to the anterior margin of tibia and pointing to the lateral malleolus. Knee extension deficit is noted as a negative value.

ROM for the ankle joint is measured with extended knee. The child is positioned in supine position. The subtalar joint is stabilized by the examinator fixating the calcaneus. The intertarsal movement is inhibited by slightly inverting the forefoot. The fixed arm of the goniometer will be parallel to the anterior margin of the tibia and the moving arm parallel to the lateral margin of the foot. 90 degree in the ankle will be noted as 0 degree. Dorsal flexion less than 0 degree will be noted as a negative value.

The two investigators will do measurements separate and blinded from each other. Data including age, sex, spastic side (right/left), Gross Motor Classification System level (GMFCS), use of orthosis and level of spasticity according to Ashworth. Level of spasticity on the spastic side will be a consensus decision by the two investigators.

Statistics Statistical power analyses calculations imply that the planned study need at least 32 children to examine 64 legs. Inter-rater reliability will be evaluated using Intra-class correlation coefficient (ICC). Limits of agreement analysis will also be used. Effect of spasticity on the reliability of pROM measurement will be evaluated comparing the ICC on the spastic leg to the non spastic leg.

Ethics The risk of causing physical harm to the research participants is considered very low. Evaluating pROM is part of regular assessment of these children. The time consumed by participating in the study might be extra compared to normal follow up but is very limited and proportional to valuable information that might be the result of the study. To minimize the pressure on families to participate, families under treatment from the researchers will primarily not be approached. Data collected will be stored in a safe way on encrypted hard drive. Personal numbers will be replaced by serial numbers and only the main researcher will have the code key.

Importance The risk of joint contracture is a major cause for concern in the growing child with cerebral palsy and something that is closely monitored by physicians and physiotherapists. Delayed diagnosis of joint contracture often leads to surgical release, a last option of treatment. The main tool for monitoring is by ROM measurements on a regular basis. Early detection of a decreasing ROM is vital for successful treatment and optimal outcome over time. The current study will add further knowledge on how ROM measurements can be interpreted and so hopefully lead to improved care for this group of children. The results will also be of importance to the research field for planning future studies and interpreting results.

ELIGIBILITY:
Inclusion Criteria: Children with hemiplegic spastic cerebral palsy -

Exclusion Criteria: Other cerebral palsy diagnoses. Surgery or botulinum toxin treatment within 3 month prior to examination.

-

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with with hemiplegic spastic cerebral palsy in the south of Sweden, Skane county.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Ankle range of motion | 2023-2024
  Goniometer measurements of ankle range of movement
Knee range of motion | 2023-2024
  Goniometer measurements of knee range of movement

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Hägglund, Study Director — Lund University
Locations (1):
- Children Habilitation Unit, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allington NJ, Leroy N, Doneux C. Ankle joint range of motion measurements in spastic cerebral palsy children: intraobserver and interobserver reliability and reproducibility of goniometry and visual estimation. J Pediatr Orthop B. 2002 Jul;11(3):236-9. doi: 10.1097/00009957-200207000-00007. PMID 12089500
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Brosseau L, Balmer S, Tousignant M, O'Sullivan JP, Goudreault C, Goudreault M, Gringras S. Intra- and intertester reliability and criterion validity of the parallelogram and universal goniometers for measuring maximum active knee flexion and extension of patients with knee restrictions. Arch Phys Med Rehabil. 2001 Mar;82(3):396-402. doi: 10.1053/apmr.2001.19250. PMID 11245764
- [Background] Ferriero G, Vercelli S, Sartorio F, Munoz Lasa S, Ilieva E, Brigatti E, Ruella C, Foti C. Reliability of a smartphone-based goniometer for knee joint goniometry. Int J Rehabil Res. 2013 Jun;36(2):146-51. doi: 10.1097/MRR.0b013e32835b8269. PMID 23196790
- [Background] Gandbhir VN, Cunha B. Goniometer. 2020 Jun 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK558985/ PMID 32644411
- [Background] Hancock GE, Hepworth T, Wembridge K. Accuracy and reliability of knee goniometry methods. J Exp Orthop. 2018 Oct 19;5(1):46. doi: 10.1186/s40634-018-0161-5. PMID 30341552
- [Background] Herrero P, Carrera P, Garcia E, Gomez-Trullen EM, Olivan-Blazquez B. Reliability of goniometric measurements in children with cerebral palsy: a comparative analysis of universal goniometer and electronic inclinometer. A pilot study. BMC Musculoskelet Disord. 2011 Jul 10;12:155. doi: 10.1186/1471-2474-12-155. PMID 21740600
- [Background] Konor MM, Morton S, Eckerson JM, Grindstaff TL. Reliability of three measures of ankle dorsiflexion range of motion. Int J Sports Phys Ther. 2012 Jun;7(3):279-87. PMID 22666642
- [Background] Martin RL, McPoil TG. Reliability of ankle goniometric measurements: a literature review. J Am Podiatr Med Assoc. 2005 Nov-Dec;95(6):564-72. doi: 10.7547/0950564. PMID 16291848
- [Background] McDowell BC, Hewitt V, Nurse A, Weston T, Baker R. The variability of goniometric measurements in ambulatory children with spastic cerebral palsy. Gait Posture. 2000 Oct;12(2):114-21. doi: 10.1016/s0966-6362(00)00068-0. PMID 10998607
- [Background] McWhirk LB, Glanzman AM. Within-session inter-rater realiability of goniometric measures in patients with spastic cerebral palsy. Pediatr Phys Ther. 2006 Winter;18(4):262-5. doi: 10.1097/01.pep.0000234960.88761.97. PMID 17108799
- See also: CPUP IS A FOLLOW-UP SURVEILLANCE PROGRAMME FOR PEOPLE WITH CEREBRAL PALSY (CP) — https://cpup.se/